CLINICAL TRIAL: NCT06288555
Title: Validation of Ipswich Touch Test for Diabetic Peripheral Neuropathy Screening in Primary Care
Status: Completed | Type: Observational
Sponsor: Ponlawat Hanchana, MD (Other Government)
Responsible Party: Sponsor-Investigator, Ponlawat Hanchana, MD, Principal Investigator, PhraPhutthabat Hospital
Organization: PhraPhutthabat Hospital (Other Government)
Other Study IDs: 020/2566
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Foot
Keywords: Diabetes mellitus; Ipswich touch test; Accuracy; Sensitivity
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patient: This study focused on a group of 274 patients with type 2 diabetes who were receiving services at Nong Khantee Subdistrict Health Promoting Hospital in Phra Phutthabat District, Saraburi Province. Participants underwent both the Ipswich touch test and the 10-g monofilament test.
  Interventions: Diagnostic Test: Ipswich touch test

INTERVENTIONS:
Diagnostic Test: Ipswich touch test — Ipswich touch test: A simple test to screen for diabetic peripheral neuropathy (DPN) by lightly touching the patient's toes with the index finger and asking them to identify which foot is touched.
  10g monofilament test: A more sensitive test to confirm DPN by applying a thin nylon fiber to different sites on the patient's feet and asking them to indicate when they feel the pressure.
  Test procedure: The patient closes their eyes and the examiner performs both tests in a specific sequence and records the results. The tests are done on healthy skin and not on wounds or calluses.
  Other Names: 10-g monofilament test

SUMMARY:
The goal of this observational study is to assess the accuracy of screening for diabetic peripheral neuropathy by comparing the Ipswich touch test with the 10-g monofilament test in patients diagnosed with type 2 diabetes.

The main question it aims to answer is:

How does the accuracy of the Ipswich Touch Test for identifying peripheral neuropathy compare to the traditional 10-g monofilament test?

Participants underwent both the Ipswich touch test and the 10-g monofilament test.

DETAILED DESCRIPTION:
BACKGROUND: Diabetic foot, a severe complication of diabetes, significantly impairs the quality of life of affected individuals. However, it can be prevented through screening for loss of protective sensation in the foot. Currently, standard screening methods still require specialized equipment and trained medical professionals.

OBJECTIVES: The aim of this study is to assess the accuracy of screening for diabetic peripheral neuropathy by comparing the Ipswich touch test with the 10-g monofilament test in patients diagnosed with type 2 diabetes.

METHODS: This diagnostic study with a cross-sectional design focused on a group of 274 patients with type 2 diabetes who were receiving services at Nong Khantee Subdistrict Health Promoting Hospital in Phra Phutthabat District, Saraburi Province. Participants underwent both the Ipswich touch test and the 10-g monofilament test. Statistical analysis included evaluating sensitivity, specificity, negative predictive value, positive predictive value, negative likelihood ratio, positive likelihood ratio, and Cohen's kappa statistic to assess the diagnostic reliability of the Ipswich touch test.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old or older, having type 2 diabetes
* being able to communicate in Thai by speaking and listening.

Exclusion Criteria:

* AIDS
* Alcoholism
* Any cancer
* Cerebrovascular disease
* Chronic foot ulcers, or having foot or toe amputation.
* Chronic kidney disease stage 4 and 5
* Cirrhosis
* Malnutrition
* Neurological disease
* Thyroid hormone deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who were receiving services at Nong Khantee Subdistrict Health Promoting Hospital(Primary care) in Phra Phutthabat District, Saraburi Province.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
The accuracy of the Ipswich touch test | 1 year
  sensitivity, specificity, negative predictive value, positive predictive value, negative likelihood ratio, and positive likelihood ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ponlawat Hanchana, MD., Principal Investigator — PhraPhutthabat Hospital
Locations (1):
- Ponlawat Hanchana, MD, Changwat Sara Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data was save inform of Microsoft excel spreadsheet and Stata file.

REFERENCES:
- [Background] International Diabetes Federation. Diabetes Facets and Figures [Internet]. Brussels: International Diabetes Federation; c2023 [updated 2023 Oct 20; cited 2023 Oct 22]. Available from: https://idf.org/about-diabetes/diabetes-facts-figures/
- [Background] Department of Disease Control. World Diabetes Day Campaign 2021: Emphasizing the importance of diabetes care to ensure widespread treatment [Internet]. Ministry of Public Health; c2021 [updated 2023 Jan 21; cited 2023 Oct 22]. Available from: https://ddc.moph.go.th/brc/news.php?news=21692&deptcode=brc
- [Background] Leelawattana R, Pratipanawatr T, Bunnag P, Kosachunhanun N, Suwanwalaikorn S, Krittiyawong S, Chetthakul T, Plengvidhya N, Benjasuratwong Y, Deerochanawong C, Mongkolsomlit S, Ngarmukos C, Rawdaree P. Thailand diabetes registry project: prevalence of vascular complications in long-standing type 2 diabetes. J Med Assoc Thai. 2006 Aug;89 Suppl 1:S54-9. PMID 17717878
- [Background] Thirapatarapong W., Srisawasdi G. Epidemiology and direct cost of diabetes related lower extremity amputations at Siriraj hospital. Journal Thai Rehabil Med 2008;18(2):65-9.
- [Background] Rerkasem K, Kosachunhanun N, Tongprasert S, Khwanngern K, Matanasarawoot A, Thongchai C, Chimplee K, Buranapin S, Chaisrisawadisuk S, Manklabruks A. The development and application of diabetic foot protocol in Chiang Mai University Hospital with an aim to reduce lower extremity amputation in Thai population: a preliminary communication. Int J Low Extrem Wounds. 2007 Mar;6(1):18-21. doi: 10.1177/1534734606298285. PMID 17344197
- [Background] Medical Research and Technology Assessment Institute. Department of Medical Services. Ministry of Public Health. Clinical Practice Guideline: Prevention and Management of Diabetic Foot Complications. Bangkok: New Thammada Printing (Thailand) Co., Ltd.; 2014.
- [Background] Moxey PW, Gogalniceanu P, Hinchliffe RJ, Loftus IM, Jones KJ, Thompson MM, Holt PJ. Lower extremity amputations--a review of global variability in incidence. Diabet Med. 2011 Oct;28(10):1144-53. doi: 10.1111/j.1464-5491.2011.03279.x. PMID 21388445
- [Background] Gibson TB, Driver VR, Wrobel JS, Christina JR, Bagalman E, DeFrancis R, Garoufalis MG, Carls GS, Gatwood J. Podiatrist care and outcomes for patients with diabetes and foot ulcer. Int Wound J. 2014 Dec;11(6):641-8. doi: 10.1111/iwj.12021. Epub 2013 Feb 4. PMID 23374540
- [Background] Thai Diabetes Society. Clinical practice guideline for diabetes 2023. Bangkok: Thai Diabetes Society; 2023. p. 165-178.
- [Background] Sudjai N. Sample size calculation for diagnostic test studies. J Med Health Sci. 2020 Aug. 31;27(2):167-82.
- [Result] Sharma S, Kerry C, Atkins H, Rayman G. The Ipswich Touch Test: a simple and novel method to screen patients with diabetes at home for increased risk of foot ulceration. Diabet Med. 2014 Sep;31(9):1100-3. doi: 10.1111/dme.12450. Epub 2014 Apr 11. PMID 24673517
- [Result] Bowling FL, Abbott CA, Harris WE, Atanasov S, Malik RA, Boulton AJ. A pocket-sized disposable device for testing the integrity of sensation in the outpatient setting. Diabet Med. 2012 Dec;29(12):1550-2. doi: 10.1111/j.1464-5491.2012.03730.x. PMID 22672290
- [Result] Dutra LMA, Moura MC, do Prado FA, De Oliveira Lima G, Melo MC, Fernandez RNM, Novaes MRCG. Is it possible to substitute the monofilament test for the Ipswich Touch Test in screening for peripheral diabetic neuropathy? Diabetol Metab Syndr. 2020 Mar 31;12:27. doi: 10.1186/s13098-020-00534-2. eCollection 2020. PMID 32266011
- [Result] Rayman G, Vas PR, Baker N, Taylor CG Jr, Gooday C, Alder AI, Donohoe M. The Ipswich Touch Test: a simple and novel method to identify inpatients with diabetes at risk of foot ulceration. Diabetes Care. 2011 Jul;34(7):1517-8. doi: 10.2337/dc11-0156. Epub 2011 May 18. PMID 21593300